CLINICAL TRIAL: NCT06829732
Title: Closed Loop Oxygen Control in INtubated Critically Ill Patients - CLOC-IN
Brief Title: Closed Loop Oxygen Control in INtubated Critically Ill Patients
Acronym: CLOC-IN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Oriol Roca, Director of Critical Care Department, Corporacion Parc Tauli
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PT_UCI_RESP1
Record Dates: First submitted 2024-01-15; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Hypoxemic Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Every patient included will be randomize to recieved both arm in different order. Every period will last for 4 h.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. closed-loop oxygen control (CLOC) (Experimental): Automatic Oxygen management sets the Oxygen control according to the patient's measured SpO2 and the operator-set SpO2 target range during 4h.
  Interventions: Device: closed-loop oxygen control (CLOC)
- 2. manual oxygen titration (MOT) (Active Comparator): Conventional oxygen manual management according to SpO2 target range set by clinician, during 4h.
  Interventions: Device: 2. manual oxygen titration (MOT)

INTERVENTIONS:
Device: closed-loop oxygen control (CLOC) — HAMILTON-C6 (Hamilton Medical, Bonaduz, Switzerland) ventilators will be used. It allows for O2 Assist software, that will be installed on all C6 ventilators before the start of this study. Automatic Oxygen management sets the Oxygen control according to the patient's measured SpO2 and the operator-set SpO2 target range. The Oxygenation controller will be activated for 4h and adjusts the Oxygen according to patient's measured SpO2.
  Arms: 1. closed-loop oxygen control (CLOC)
Device: 2. manual oxygen titration (MOT) — O2 will be manually set according to SpO2 target during a 4h period.
  Arms: 2. manual oxygen titration (MOT)

SUMMARY:
The deleterious effects of alveolar hyperoxia and (severe) hyperoxaemia are well described. Achieving safe and efficient oxygenation may be challenging. The hypothesis of the present study is that closed-loop oxygen control in intubated and mechanically ventilated critically ill patients improves oxygen administration compared with standard manual oxygen titrations. A single-blind, randomised crossover clinical trial assessing the efficacy and safety of the use of a closed-loop oxygen control versus manual oxygen titration in patients receiving mechanical ventilation has been designed. Patients will be randomised to receive first either closed-loop oxygen control (CLOC) or manual oxygen titration (MOT). The percentage of time spent in optimal and sub-optimal SpO2 (oxygen saturation by pulse oximetry) ranges will be calculated for each period.

DETAILED DESCRIPTION:
The deleterious effects of alveolar hyperoxia and (severe) hyperoxaemia are well described. A safe and efficient oxygenation should be achieved. However, from a practical point of view, this may require frequent manual adjustments of the inspired oxygen, which might be unfeasible, especially in high-demand periods. Several automatic oxygen systems have been tested in non-intubated patients. The hypothesis of the present study is that closed-loop oxygen control in intubated and mechanically ventilated critically ill patients improves oxygen administration compared with standard manual oxygen titrations. Thus, the objective of the study is to compare the percentage of time spent in a predefined optimal SpO2 range between closed-loop oxygen control and manual oxygen titration.

A single-blind, randomised crossover clinical trial assessing the efficacy and safety of the use of a closed-loop oxygen control versus manual oxygen titration in patients receiving mechanical ventilation has been designed. Once included, patients will be randomised to receive first either closed-loop oxygen control (CLOC) or manual oxygen titration (MOT). Every period will last for 4h. Clinical and respiratory variables will be recorded. A memory box will be connected to the patient's ventilator. This device will record ventilator parameters, including FiO2 and SpO2. To assess the outcome, the percentage of time spent in optimal and sub-optimal SpO2 ranges will be calculated for each period.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU who are expected to require invasive mechanical ventilation for at least 8 hours and are expected to stay respiratory stable´ in the upcoming 8 hours.
* Acute respiratory failure with PaO2/FiO2 <300 with FiO2 ≥ 0.4 at inclusion
* Age older than 18 years old.
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation.

Exclusion Criteria:

* Low quality on the SpO2 measurement using finger and ear sensor (quality index <60%).
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h.
* Severe acidosis (pH ≤ 7.30).
* Chronic or acute dyshemoglobinemia: methemoglobin, CO poisoning, sickle cell disease.
* Patient under guardianship or deprived of liberties.
* Impossibility to give informed consent by both patient and family (i.e. language barrier).
* Patient included in another interventional research study under consent with similar outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy outcome: | Hour 1 to 4
  To compare the percentage of time spent in a predefined optimal SpO2 (oxygen saturation by pulse oximetry) range between closed-loop oxygen control and manual oxygen titration

SECONDARY OUTCOMES:
Percentage of time with SpO2 (oxygen saturation by pulse oximetry) in sub-optimal ranges | Hour 1 to 4
  To compare the percentage of time with SpO2 in sub-optimal ranges, above and below the optimal range, during closed-loop oxygen control and manual oxygen titration
Percentage of time with SpO2 (oxygen saturation by pulse oximetry) out of range | Hour 1 to 4
  To compare the percentage of time with SpO2 out of range, above and below the optimal and sub-optimal range.
Number of manual adjustments | Hour 1 to 4
  To compare the number of manual adjustments
Mean SpO2/FiO2 (oxygen saturation by pulse oximetry to fraction of inspired oxygen ratio) between the two methods | Hour 1 to 4
  To compare the mean SpO2/FiO2 between the two methods of oxygen titration
Mean FiO2 (fraction of inspired oxygen) between the two methods of oxygen titration | Hour 1 to 4
  To compare the mean FiO2 between the two methods of oxygen titration
Time with FiO2 (fraction of inspired oxygen) below 40% | Hour 1 to 4
  To compare the percentage of time with FiO2 below 40%
Time with FiO2 (fraction of inspired oxygen) above 60% | Hour 1 to 4
  To compare the percentage of time with FiO2 above 60%
Time with FiO2 (fraction of inspired oxygen) at 100% | Hour 1 to 4
  To compare the percentage of time with FiO2 at 100%
SpO2 (oxygen saturation by pulse oximetry) below 88 and 85%. | Hour 1 to 4
  To compare the percentage of time with SpO2 below 88 and 85%.
SpO2 (oxygen saturation by pulse oximetry) below 88 and 85% (Event > 10s and 60 s) | Hour 1 to 4
  To compare the number of events with SpO2 below 88 and 85% (Event > 10s and 60 s)
Number of alarms | Hour 1 to 4
  To compare the number of alarms
Time with SpO2 (oxygen saturation by pulse oximetry) signal available. | Hour 1 to 4
  To compare the percentage of time with SpO2 signal available.
Total amount of oxygen used | Hour 1 to 4
  To compare the total amount of oxygen used (in L)

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Tauli Hospital Universitary, Sabadell, Barcelona, Spain